CLINICAL TRIAL: NCT03461315
Title: "COMPARATIVE STUDY OF TWO MODELS OF PREVENTIVE HOME VISITS "
Brief Title: Comparative Study Between Two Models of Home Care.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Badalona Serveis Assistencials (Other)
Collaborators: Rosa Maria Sequera Requero (Unknown); Sebastià J. Santaeugènia González (Unknown); Francisco José Tarazona Santabalbina (Unknown)
Responsible Party: Principal Investigator, Carolina Burgos Diez, Family physician, Badalona Serveis Assistencials
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: P17/121
Record Dates: First submitted 2018-03-05; First posted 2018-03-12 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2018-03

CONDITIONS: Managed Care Program; Home Care
Keywords: home care; primary care; preventive home visits

STUDY DESIGN:
Intervention Model Description: Quasi-experimental study .
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Mode (No Intervention): Traditional Model: Team That Cares for the Rest of the Community
- Study Model (Experimental): Study Model:Team Dedicated Exclusively to the Home Patient
  Interventions: Other: Functional assistance model

INTERVENTIONS:
Other: Functional assistance model — Preventive home visits carried out by a Team Dedicated Exclusively to the Home Patient.
  Arms: Study Model

SUMMARY:
Home care is the assistance provided at home to those who can not travel to their Health Center. There are multiple studies on models of home care and many discrepancies about the impact that preventive home visits can have. Hypothesis: home care is expected to be better if performed by a team dedicated exclusively to the home patient, than to the traditional model, where the patient is assisted by the team that cares for the rest of the community.

Goals:

Main: determine the difference in median cumulative days of hospital admission in 12 months.

Secondaries:

* results in health
* in health experience in efficiency Methodology: Quasi-experimental study of two years duration. All the subjects included in the Home Care Program and that meet the inclusion and exclusion criteria are studied. The care team will provide the informed consent and information sheet to the patient and clinical scales at the beginning and end of the study. Researchers will be responsible for the collection of data that they will anonymize and guard. Statistical analysis: The analyzes will be calculated with the statistical package SPSS version 21 Expected results: hospital admissions (25%) and cumulative days by admission and patient by 65% are expected to improve in the model under study. Applicability and relevance: the trend towards a greater aging of the population makes it necessary to study models of care that allow us to detect which can be beneficial to the population and feasible in our current context.

DETAILED DESCRIPTION:
Our purpose will be to compare 2 models of home care corresponding to 2

Primary Care Centers (EAP):

* Model integrated (EAP Gran Sol), traditional, continuity, made by the UBA with care of the home patient by the usual care team (family physician and nurse)
* Model functional (EAP Apenins), based on the internal reorganization of the EAP: equipment specific home care program composed of family physician and nurse, with dedication exclusively to Preventive home visits, with training aimed at excellence in the Management of fragile patients with pluripathology and palliative care.

HYPOTHESIS. A care group dedicated exclusively to the ATDOM patient with what it entails in dedication of time and specific knowledge could get better results in health, optimize health resources and at the same time achieve greater satisfaction and quality of life to these patients. That is why our hypothesis will be that it is expected that the patient's global assistance attended from Primary Care in your home is better if it is performed by a Primary Care team trained for it with exclusive dedication to this type of patient, that, with the traditional model, where the patient that is attended at home is assisted by the clinical team that serves the rest of the community.

OBJECTIVES Main objective The main objective will be the comparison of the two models of home care in Primary care previously described by the difference in the average number of days hospitalized for 12 months among the people served in an integrated model of home care and among those served in a functional model. 3.2 Secondary objectives We will analyze them under a triple vision AIM, triple goal, better health, better care, lower costs, -effectiveness, efficiency and experience in people's health-

* Results in health: comparison in mortality at 12 months and integral geriatric assessment.
* Results in experience in health care and quality of life:

Comparison of both models in terms of self-perception in patients' health included in the preventive home care program, the patient's experience in attention to their health and overload of the caregiver.

-Results in efficiency and resource utilization: comparison in professional assistance, consumption of intermediate resources, consumption of social products, quality in the prescription.

METHODOLOGY OF THE STUDY.

* Design of the study. It is a quasi-experimental study of 2 population samples. The group of study is composed of the sample of subjects treated with the home care model exclusive and expert. The control group is made up of the subjects that are treated with the model of traditional home care. The study is expected to have a duration of 2 years that will be the time of follow-up of each participant, being able present the possibility of doing later substudies.
* Population under study. Justification of the choice of the comparator. The integrated model of home care that is implemented in EAP Gran Sol is compared with the proposed new functional model that includes a team of family doctor and nurse dedicated exclusively to patient care included in the home care program and who have received specific training. This intervention has been carried out in EAP Apenins since 2013.

To the subjects of this obtained sample, a telephone call will be made inviting them to participate in the study, agreeing a visit by the doctor or nurse responsible for the patient and the subject of the project will be informed. In the agreed view, will give the informed consent and the information sheet to the patient. Once signed in informed consent by the subject or in case of patients with deterioration cognitive, by the caregiver, the self-administered scales EuroQOL and IEXPACto the patient, in the case of patients with cognitive impairment, at caregiver and the Zarit questionnaire to the main caregiver so that complete They will be given an envelope to enter the completed scales that will be delivered closed to the healthcare professional. Fragility will be measured with instrument of Gérontopole at that time. These scales will be redelivered the patient and the caregiver at the end of the study, after 2 years, with the same methodology.

It is considered inevitable that professionals know how to measure themselves since they have their collaboration for the delivery of informed consent and information sheet to patient and the EuroQol, IEXPAC and Zarit scales and calculation of fragility index.

There will be 2 training sessions for healthcare professionals on the project of the study and the use of the scales they will deliver. Losses of selection of the sample are considered to the subjects or main caregivers, in the case of subjects with cognitive impairment, who do not sign informed consent.

Every 6 months the researchers will contact the subjects by telephone participants of the study (each of their Primary Care Center) and on that call will proceed to question about possible admission to private hospitals, stay in day centers or answer questions or provide information about the study. Study groups.

They are the following:

A control group of patients included in the Home Care program of the ABS Gran Sol where11 healthcare teams work with 241 patients in total in the Home care program (date December 2016) And a study group, of patients included in the Home Care program of ABS Apenins, the which have a healthcare team that works exclusively for home care with 113 patients (date December 2016) Study sample. Patients will be included who are in the Home care program and who comply with the Inclusion and exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

-Patients of 65 or more years, with or without cognitive impairment, that during the period of recruitment are new or existing users in a home care program long duration of the centers participants.

Exclusion Criteria:

* the patients who have a life expectancy of less than 1 month, considering that provides information for this study and may not be appropriate for the patient and the operating system relatives
* patients with Pfeiffer index mayor or equal to 5 without primary caregiver or with a partial caregiver, since we consider that with moderate cognitive impairment or severe will not be able to answer self-administered questionnaires.
* the patients included in the home care program for the performance of cures or treatments that 3 months (Transient home care Program).
* the patients who have been in the home care program for less than 1 month at the time of their recruitment, since we believe that there has not yet been time to carry out a comprehensive assessment of the patient.
* the patients included in the home care program who are not registered in Badalona because they are temporarily in the home of a family member.
* the patients included in the home care Program due to the existence of barriers architectures to go to the Primary Care Center.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 354 (Estimated)
Dates: Start 2018-04-01 (Estimated); Primary Completion 2018-07-01 (Estimated); Study Completion 2020-04-01 (Estimated)

PRIMARY OUTCOMES:
difference in the average of days hospitalized for 12 months among the people served in an integrated model of home care and among those served in a functional model. | 2 years

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Burgos-Diez C, Sequera-Requero RM, Tarazona-Santabalbina FJ, Contel-Segura JC, Monzo-Planella M, Santaeugenia-Gonzalez SJ. Study protocol of a quasi-experimental trial to compare two models of home care for older people in the primary setting. BMC Geriatr. 2020 Mar 12;20(1):101. doi: 10.1186/s12877-020-1497-0. PMID 32164542